CLINICAL TRIAL: NCT01243567
Title: Safety and Efficacy of Bimatoprost/Timolol Fixed Combination Versus Latanoprost in Patients With Open-Angle Glaucoma Who Have Never Been Treated
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAF-AGN-OPH-GLA-010; 2009-012799-28 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Bimatoprost; Timolol; Ganfort; Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimatoprost 0.03%/timolol 0.5% combination ophthalmic solution (Active Comparator): Bimatoprost 0.03%/timolol 0.5% combination ophthalmic solution (GANfort®) administered to each eye requiring treatment, once daily in the evening for 3 months.
  Interventions: Drug: bimatoprost 0.03%/timolol 0.5% combination ophthalmic solution
- latanoprost 0.005% ophthalmic solution (Active Comparator): Latanoprost 0.005% ophthalmic solution (Xalatan®) administered to each eye requiring treatment, once daily in the evening for 3 months.
  Interventions: Drug: latanoprost 0.005% ophthalmic solution

INTERVENTIONS:
Drug: bimatoprost 0.03%/timolol 0.5% combination ophthalmic solution — Bimatoprost 0.03%/timolol 0.5% combination ophthalmic solution (GANfort®) administered to each eye requiring treatment, once daily in the evening for 3 months.
  Other Names: GANFort®
  Arms: bimatoprost 0.03%/timolol 0.5% combination ophthalmic solution
Drug: latanoprost 0.005% ophthalmic solution — Latanoprost 0.005% ophthalmic solution (Xalatan®) administered to each eye requiring treatment, once daily in the evening for 3 months.
  Other Names: Xalatan®
  Arms: latanoprost 0.005% ophthalmic solution

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost/timolol fixed combination (GANfort®) versus latanoprost (Xalatan®) in patients with open-angle glaucoma who have never been previously treated and are at high risk for progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma that has never been treated
* Visual Acuity 20/60 or better in each eye

Exclusion Criteria:

* Eye surgery within 3 months
* Any refractive eye surgery
* Contraindication to beta-adrenoceptor antagonist therapy (eg, chronic obstructive pulmonary disease [COPD], bronchial asthma, sinus bradycardia, heart block, history of severe myocardial infarction [heart attack])
* Eye inflammation or eye infection within 3 months
* Eye trauma within 6 months
* Oral, injectable, or topical ophthalmic steroids within 21 days or anticipated use during study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2012-02-14 (Actual); Study Completion 2012-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Coimbra, Portugal
- Madrid, Spain

REFERENCES:
- [Background] Gutierrez-Diaz E, Silva Cotta J, Munoz-Negrete FJ, Gutierrez-Ortiz C, Morgan-Warren RJ, Maltman J. Bimatoprost/timolol fixed combination versus latanoprost in treatment-naive glaucoma patients at high risk of progression: a pilot study. Clin Ophthalmol. 2014 Apr 10;8:725-32. doi: 10.2147/OPTH.S56735. eCollection 2014. PMID 24748767

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution
Started | 43 | 38
Completed | 42 | 38
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution | Total
Number analyzed (Participants) | 43 | 38 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (10.24) | 63.1 (13.72) | 64.6 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. For each patient, the IOP is the average of the two eyes. The average IOP is the average of the 08:00, 12:00 and 16:00 hour time points at each visit for each patient. A negative number change from Baseline indicates a reduction in average IOP (improvement).
Time Frame: Baseline, Month 3
Population: Intent to Treat: all randomized patients.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution
Number analyzed (Participants) | 43 | 38
Millimeters of Mercury (mmHg)
  Baseline | 28.4 (3.35) | 28.5 (2.57)
  Change from Baseline at Month 3 | -13.5 (4.48) | -11.4 (3.19)

2. Secondary Outcome: Change From Baseline IOP
Description: IOP is a measurement of the fluid pressure inside the eye. For each patient, the IOP is the average of the two eyes. IOP is recorded at the 08:00 (8:00 am), 12:00 (noon) and 16:00 (4:00 pm) hour time points for each patient at each visit. A negative number change from Baseline indicates a reduction in IOP (improvement).
Time Frame: Baseline, Month 3
Population: Intent to Treat: all randomized patients.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution
Number analyzed (Participants) | 43 | 38
Millimeters of Mercury (mmHg)
  Baseline-08:00 | 29.7 (2.97) | 29.6 (2.93)
  Baseline-12:00 | 28.7 (4.46) | 29.0 (2.60)
  Baseline-16:00 | 26.8 (4.01) | 26.8 (3.73)
  Change from Baseline at Month 3-08:00 | -14.6 (4.04) | -12.3 (3.64)
  Change from Baseline at Month 3-12:00 | -13.6 (5.50) | -11.8 (3.14)
  Change from Baseline at Month 3-16:00 | -12.4 (5.16) | -10.3 (4.24)

3. Secondary Outcome: Percentage of Patients Reaching a Predefined Target Pressure Threshold
Description: IOP is a measurement of the fluid pressure inside the eye. For each patient, the IOP is the average of the two eyes. The predefined target pressure thresholds are at least a 20%, 30%, 40%, and 50% reduction in IOP from baseline.
Time Frame: Baseline, Month 3
Population: Intent to Treat: all randomized patients.
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution
Number analyzed (Participants) | 43 | 38
Percentage of Patients
  Decrease of at Least 20% | 97.7 | 100.0
  Decrease of at Least 30% | 90.7 | 86.8
  Decrease of at Least 40% | 74.4 | 47.4
  Decrease of at Least 50% | 46.5 | 15.8

4. Secondary Outcome: Absolute Difference Between Patient's Highest IOP Reading at Baseline (Day 0) and the Corresponding IOP Reading
Description: IOP is a measurement of the fluid pressure inside the eye. Two or three measurements of IOP are taken for each eye at each time point. The highest IOP values between the two eyes for each patient at each time point are used to calculate the absolute difference.
Time Frame: Baseline, Month 3
Population: Intent to Treat: all randomized patients.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution
Number analyzed (Participants) | 43 | 38
Millimeters of Mercury (mmHg)
  Baseline | 30.4 (3.19) | 30.3 (2.54)
  Absolute Difference at Month 3 | -15.3 (4.44) | -12.9 (3.82)

5. Secondary Outcome: Absolute Difference Between Patient's Lowest IOP Reading at Baseline (Day 0) and the Corresponding IOP Reading
Description: IOP is a measurement of the fluid pressure inside the eye. Two or three measurements of IOP are taken for each eye at each time point. The lowest IOP values between the two eyes for each patient at each time point are used to calculate the absolute difference.
Time Frame: Baseline, Month 3
Population: Intent to Treat: all randomized patients.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution
Number analyzed (Participants) | 43 | 38
Millimeters of Mercury (mmHg)
  Baseline | 26.2 (4.04) | 26.5 (3.44)
  Absolute Difference at Month 3 | -11.8 (5.23) | -9.9 (3.71)

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution | Latanoprost 0.005% Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/38
Other Adverse Events (participants affected / at risk) | 9/43 | 10/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution (N=43) | Latanoprost 0.005% Ophthalmic Solution (N=38)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03%/Timolol 0.5% Combination Ophthalmic Solution (N=43) | Latanoprost 0.005% Ophthalmic Solution (N=38)
Ocular Hyperaemia (Eye disorders) | 7 | 4
Blepharitis (Eye disorders) | 1 | 2
Conjunctival Hyperaemia (Eye disorders) | 1 | 2
Foreign Body Sensation in Eyes (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.